CLINICAL TRIAL: NCT07108621
Title: Eight Weeks of Low Dose hCG Priming in Women With Diminished Ovarian Reserve Undergoing IVF/ICSI - a Randomized Controlled Trial
Brief Title: hCG Priming in Women With Diminished Ovarian Reserve
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kristine Loessl (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Copenhagen University Hospital at Herlev (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristine Loessl, Associate professor, Ph.D., MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-521234-28; 2025-521234-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-11; First posted 2025-08-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Infertility, Female; Ovarian Reserve; In Vitro Fertilization (IVF)
Keywords: hCG priming; Androgen priming; Diminished ovarian reserve; In vitro fertilization (IVF); Controlled ovarian stimulation
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hCG Priming (Experimental): Women in the experimental group will undergo the following treatment in order:
  A standard IVF/ICSI cycle (ICSI I): A standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and a GnRH antagonist (Ganirelix 0.25 mg) from stimulation day 5-6 followed by blastocyst culture and a freeze-all strategy.
  Priming period: hCG priming 260 IU once daily for two menstrual cycles (approximately 8 weeks).
  A standard IVF/ICSI cycle (ICSI I): A standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and a GnRH antagonist (Ganirelix 0.25 mg) from stimulation day 5-6 followed by blastocyst culture and a single blastocyst transfer at day 5.
  Interventions: Drug: Choriongonadotropin alfa (hCG)
- Placebo (Placebo Comparator): Women in the placebo group will undergo the following treatment in order:
  A standard IVF/ICSI cycle (ICSI I): A standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and a GnRH antagonist (Ganirelix 0.25 mg) from stimulation day 5-6 followed by blastocyst culture and a freeze-all strategy.
  Priming period: Placebo (isotone NaCl) injections once daily for two menstrual cycles (approximately 8 weeks).
  A standard IVF/ICSI cycle (ICSI I): A standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and a GnRH antagonist (Ganirelix 0.25 mg) from stimulation day 5-6 followed by blastocyst culture and a single blastocyst transfer at day 5.
  Interventions: Drug: Isotonic NaCl (Placebo)

INTERVENTIONS:
Drug: Choriongonadotropin alfa (hCG) — hCG 260 IU once daily for two menstrual cycles (aproximately 8 weeks) prior til standard IVF/ICSI.
  Arms: hCG Priming
Drug: Isotonic NaCl (Placebo) — Placebo priming (isotone NaCl) once daily for two menstrual cycles (approximately 8 weeks) prior to standard IVF/ICSI.
  Arms: Placebo

SUMMARY:
The aim of this randomized controlled trial is to further examine the possible effects of low dose human chorionic gonadotropin (hCG) priming for eight weeks in women with diminished ovarian reserve (DOR) undergoing in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI). The investigators want to retest the findings of our first study in an identical paired design (NCT04643925), as an increase of 1.5 in mean number of oocytes retrieved is clinically relevant. To incorporate the strengths of a randomized controlled trial design, women will be randomized after their first ICSI treatment to receive either hCG or placebo in a double-blinded design during an eight-week priming period preceding their second ICSI treatment. The primary outcome is the number of oocytes retrieved in the second ICSI treatment.

DETAILED DESCRIPTION:
This randomized, double-blinded, placebo-controlled trial investigates whether eight weeks of low-dose hCG (LH activity) can produce a local intra-ovarian androgen priming and stimulate theca cell androgen production and improve oocyte yield during IVF/ICSI in women with diminished ovarian reserve (DOR).

The study is conducted at four public fertility clinics in Denmark: The Fertility Clinic at Copenhagen University Hospital, Rigshospitalet, the Fertility Clinic at Odense University Hospital, the Fertility Clinic at Hvidovre Hospital and the Fertility Clinic at Herlev Hospital.

Eligible women with DOR fulfilling the inclusion criteria and none of the exclusion criteria and with an indication for IVF/ICSI are enrolled. Women can participate only once.

Participating women will undergo two identical ICSI cycles, ICSI I and ICSI II, separated by an eight-week priming period with either daily low dose hCG-injections (260 IU) or placebo-injections (NaCl) according to randomization. Eight weeks of hCG/placebo priming corresponds to two natural menstrual cycles. A freeze-all strategy is applied in the first ICSI treatment.

Both ICSI cycles follow a fixed GnRH-antagonist protocol with of 300 IU rFSH initiated from cd 2-3 and the GnRH antagonist (Ganirelix 0.25 mg) from stimulation day 5-6. The patients undergo routine transvaginal ultrasound scans on cd 2/3, and per standard clinical practice until the day of ovulation trigger. Ovulation trigger by 6500 IU hCG sc is planned at 10 pm according to standard clinical practice. Oocyte retrieval will be done ~36 hours after ovulation trigger. ICSI will be used as fertilization method.

If no dominant/pre-ovulatory follicles are seen after 21 days of stimulation, the cycle is cancelled, but participants continue in the study.

In ICSI I, all embryos are cultured to the blastocyst stage and vitrification is performed on day 5/6 (Gardner score ≥3CC or 2AB/BA/BB). In ICSI II, single fresh blastocyst transfer is performed on day 5 after oocyte retrieval if criteria are met (Gardner score ≥3CC or 2AB/BA/BB). Surplus blastocysts will be vitrified on day 5/6 (Garner score ≥3CC or 2AB/BA/BB). If only day 6 blastocysts are available, freeze-all and postponed frozen embryo transfer will be planned.

Patients with a body weight <60 kg are instructed to take the study (hCG- or placebo) injections every second day according to experience from our previous study.

The priming period constitutes of two menstrual cycles of around 28 days each, and thus the priming period is approximately eight weeks in total, however, this duration may be extended for one menstrual cycle in the event of important patient-related or clinical issues or other unforeseen circumstances.

Comprehensive records of medication dispensing, and return will be kept to ensure accurate accountability.

Monitoring and data collection:

Transvaginal ultrasonography TVUS is performed at cycle day 2-3 and on trigger day in both ICSI I and ICSI II, and twice during the priming period to assess follicle count and size and endometrial thickness (mm), appearance (triple layered (yes/no) and density (hypo-, iso- or hyperdense).

Blood samples Blood samples will be drawn during ICSI I and ICSI II (on cd 2-3, on the day of ovulation trigger, and on the day of oocyte retrieval) where the following reproductive hormones will be measured: inhibin B, LH, FSH, estradiol, progesterone, 17-OH-progesterone, testosterone, androstenedione, and DHEAS. Additionally, AMH will be measured on cd 2-3 of ICSI I and ICSI II.

Additionally, a full blood sample will be kept in a research biobank for DNA analysis for deeper understanding of genetic reasons of DOR.

During the priming period, blood samples will be drawn at two times at the beginning of each menstrual cycle for measurements of reproductive hormones as mentioned above. In addition, two blood samples are collected during the priming period for the research biobank. These samples will be used for batch analysis of hCG levels after study completion to confirm patient compliance.

Additional treatment and interventions for patients included at Copenhagen University Hospital Rigshospitalet:

During the priming period of the second menstruation, the patients will undergo follicle aspiration, if possible, of unstimulated antral follicles to collect follicular fluid and granulosa cells. The follicular fluid and granulosa cells from each patient will be stored in a research biobank for batch analyses of reproductive hormones after study completion. The granulosa cells will be examined for androgen and FSH receptor expression and protein levels.

Treatment related data are collected. Further, the following data will be collected from patient files: female age, weight, height, BMI, fresh cycle number, days of stimulation, total rFSH dose, number of oocytes retrieved, number of metaphase II (MII) oocytes retrieved, fertilization rate, number and quality of day 2 embryos, number and quality of blastocysts and number of vitrified embryos/blastocysts, pregnancy and miscarriage rate after blastocyst transfer with blastocysts from ICSI II or postponed transfers from ICSI I.

Data will be transferred to an online eCRF; REDCap. The REDCap database has a complete audit trail and is based on anonymous subject identification numbers used in the trial. Data are backed up daily and stored on a server located in a locked facility in Denmark.

Statistics

Sample size calculation:

In our recently published paper on hCG priming investigated in a paired study design, the mean number (standard deviation (SD)) of oocytes retrieved was 3.2 (1.7) in the Control ICSI cycle and 4.7 (2.8) after eight weeks hCG priming. A sample size calculation using The POWER Procedure for a two-Sample t-test with Unequal Variances at a significance level of 0.05 showed that a total sample size of 78 women (39 in each group) will ensure a power of 80% or likely higher since baseline-adjustment usually leads to a substantial power gain, hence a total of 80 women will be included and randomized. Dropouts will be replaced until a total of 80 women have completed the study.

Statistical analyses:

Analyses will be performed in the per protocol population including all women completing ICSI I, the priming period, and ICSI II without any major protocol violations.

Since the primary outcome is an objective, quantifiable number that is routinely and always assessed and recorded as part of standard fertility treatment, the investigators expect study withdrawal and other violations to be limited and due to non-critical, random reasons. The total number of participants who are not per protocol will be reported, along with overall reasons for violations when available (e.g. difficulties in taking the trial medication, or personal reasons). Descriptive tables will be made to compare the characteristics of the women who are per protocol with the protocol violators and in case differential patterns occur between the randomisation groups, sensitivity analyses will be made to adjusting for potential confounders.

Spurious or implausible data points will be assessed on a case-by-case basis and excluded from the analysis if determined to be incorrect and not supported by clinical context.

The effect of hCG-priming vs placebo on the primary outcome, number of retrieved oocytes, will be evaluated using a constrained linear mixed model including period (ICSI I vs ICSI II) and the constrained treatment-period interaction as fixed effects and an unstructured covariance to account for repeated measurements on each woman. A two-sided p-value < 0.05 will be considered statistically significant for the primary analysis.

Quantitative secondary or exploratory outcomes will be analysed using a similar linear mixed model. All hormone concentrations will be log-transformed prior to analysis due to anticipated skewness. Count data will be compared between the treatments using constrained generalized estimating equations (GEE) with a log-link and an unstructured working covariance. Binary outcomes will be compared between the treatments using the Chi-Square Test. The p-values from the secondary analyses will be adjusted for multiple testing using the method of Benjamini and Hochberg which controls the false discovery rate. An adjusted p-values < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 (both inclusive)
* Regular menstrual cycle (23-35 days)
* 1.-5. IVF/ICSI cycle at inclusion
* AMH < 6.29 pmol/L (Elecsys® AMH assay)

Exclusion Criteria:

* Uterine malformations or hydrosalpinx
* Submucosal uterine myomas
* Uterine polyps
* Allergy to standard IVF/ICSI medication
* Endometriosis stage III-IV
* Preimplantation genetic testing
* Testicular sperm aspiration/extraction
* Ovarian enlargement or cysts (other than normally occurring corpora luteae)
* Gynaecological haemorrhages of unknown aetiology
* Known severe comorbidity*

  * i.e., Insulin dependent diabetes mellitus, non-insulin dependent diabetes mellitus, gastrointestinal, cardiovascular, thromboembolic (including active thromboembolic disorders), pulmonary, liver or kidney diseases, HIV or Hepatitis B/C, dysregulated thyroid disease, tumors of the hypothalamus or pituitary gland or ovarian, uterine, or mammary carcinoma.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | Through study completion, an average of 4 months
  The number of oocytes retrieved in the ICSI II treatment performed after hCG priming/placebo

SECONDARY OUTCOMES:
Number of mature oocytes | Through study completion, an average of 4 months
  Number of MII oocytes retrieved in the ICSI II treatment performed after hCG priming/placebo

OTHER OUTCOMES:
Antral follicle count | Through study completion, an average of 4 months
  Antral follicle count (2-9 mm) at cd 2-3
AMH | Through study completion, an average of 4 months
  AMH at cd 2-3
Number of pre-ovulatory follicles >16 mm | Through study completion, an average of 4 months
  Number of pre-ovulatory follicles >16 mm on trigger day
Number of follicles on hCG trigger day | Through study completion, an average of 4 months
  Number of follicles >14 mm and ≥12 mm ≥10 mm and <10 mm on hCG trigger day
Number of fertilized eggs | Through study completion, an average of 4 months
  Number of fertilized eggs (2 pronuclei)
Number of day 2 embryos | Through study completion, an average of 4 months
  Number of cleaved day 2 embryos (≥2-cell stage)
Number of good quality day 2 embryos | Through study completion, an average of 4 months
  A good quality day 2 embryo is defined as: 2-6 cells, < 20% fragmentation, cell size according to cell number, no multinucleation
Number of top-quality day 2 embryos | Through study completion, an average of 4 months
  A top-quality day 2 embryo is defined as: four cells < 20% fragmentation, equal cell size, no multinucleation
Number of blastocysts | Through study completion, an average of 4 months
  Number of blastocysts (Gardner score 1-6)
Number of good quality blastocysts day 5/6 | Through study completion, an average of 4 months
  Gardner score ≥3BB day 5 or ≥4BB day 6
Number of vitrified embryos/blastocysts | Through study completion, an average of 4 months
Total number of transferred or vitrified blastocysts | Through study completion, an average of 4 months
The number of cancelled cycles and the reasons for cancellation | Through study completion, an average of 4 months
Serum and follicular fluid hormone levels | Through study completion, an average of 4 months
  Hormone levels at predefined time-points: AMH (pmol/l), inhibin b (ng/ml), estradiol (nmol/l), progesterone (nmol/l), 17-OH-progesterone (nmol/l), LH (IU/l), FSH (IU/l), testosterone (nmol/l), androstenedione (nmol/l), hCG (IU/l)
Granulosa cell FSH, LH, and androgen receptor expression | Within 1 year of study completion
Pregnancy and live birth rates | Within 1 year of study completion
  Pregnancy and live birth rates per randomised woman.
Follicular Output Rate | Through study completion, an average of 4 months
  Follicular output rate (FORT) = pre-ovulatory follicle count (>16 (≥14/12/10) mm) at trigger day/antral follicle count at baseline (2-9 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Department of Gynaecology, Fertility and Obstetrics, Copenhagen University Hosital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
On request, the study protocol and unidentifiable individual participant data, including baseline characteristics (e.g. age, BMI, AMH, infertility and medical history), primary and secondary outcome measures, and relevant laboratory results collected during the trial, may be shared with research groups or publishers with relevant aims and a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Data will be available starting 3 months after trial completion. Data will remain available for up to 25 years after study completion, in accordance with EU and Danish regulatory requirements for clinical trials involving medicinal products.
Access Criteria: Approvals by necessary ethic committees and the Danish Data Protection Agency will be needed before sharing of data. All costs for data sharing will be covered by the party requesting the data. Data cannot be shared with research groups working on overlapping primary and secondary outcomes without prior discussion and agreement to avoid duplication of work. Requests for such use will be considered on a case-by-case basis.
  To gain access, data requestors will need to sign a data sharing agreement. Proposals of data sharing should be directed to kristine.loessl@regionh.dk.

REFERENCES:
- [Background] Friis Wang N, Bogstad JW, Pors SE, Petersen MR, Pinborg A, Yding Andersen C, Lossl K. Eight weeks of androgen priming by daily low-dose hCG injections before ICSI treatment in women with low ovarian reserve. Hum Reprod. 2023 Apr 3;38(4):716-725. doi: 10.1093/humrep/dead012. PMID 36721920